CLINICAL TRIAL: NCT04916756
Title: A Prospective Pilot Study to Explore Efficacy and Safety of Baricitinib in Active Primary Sjogren's Syndrome Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH-ZS-2497
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's Syndrome; JAK inhibitor; baricitinib; ESSDAI
MeSH Terms: conditions — Sjogren's Syndrome | interventions — baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- baricitinib 2mg per day (Experimental)
  Interventions: Drug: Baricitinib 2 MG

INTERVENTIONS:
Drug: Baricitinib 2 MG — baricitinib 2mg per day for 24 weeks

SUMMARY:
Primary Sjogren's syndrome (pSS) is a systemic autoimmune disease characterized by dysfunction of the exocrine glands, which results in sicca symptoms in affected patients. JAK/STAT signaling pathway is activated and playing as a key pathway in the differentiation and activation of many lymphocytes, so that affect the pathogenesis of many autoimmune diseases including pSS. JAK inhibitors have also been widely used in the treatment of rheumatoid arthritis and other autoimmune diseases.

Some studies have confirmed that JAK/STAT pathway is activated in patients with pSS, and JAK inhibitor may be effective for pSS. Filgotinib, the selective JAK1 inhibitor, is one of the "secondary generation" JAK inhibitors developed these years. Lee et al. found that filgotinib suppressed the IFN-induced transcription of differentially expressed genes and BAFF in human primary salivary gland epithelial cells. In addition, filgotinib-treated mice exhibited increased salivary flow rates and marked reductions in the lymphocytic infiltration of SGs, indicating that JAK inhibitors may be a novel therapeutic approach for pSS. A randomized phase 2 study is currently in progress to assess the safety and efficacy of filgotinib in adult subjects with active Sjogren's syndrome. So far, there is no evidence of the safety and efficacy of baricitinib in patients with pSS.

Baricitinib, an oral inhibitor of JAK1/JAK2, was the second JAK inhibitor approved for clinical use in RA. It has been approved for the treatment for moderate to severe active RA in adult patients who have responded inadequately to, or are intolerant to, one or more disease-modifying anti-rheumatic drugs (DMARDs). The efficacy and safety of baricitinib in RA have been extensively evaluated in pre-clinical animal models of arthritis, as well as in clinical studies. There are also some reports of baricitinib used in other autoimmune diseases, such as systemic lupus erythematosus, dermatomyositis and PMR/GCA. In a double-blind, multicenter, randomized, placebo-controlled, 24-week phase 2 study across 11 countries, baricitinib treatment at a dose of 4 mg dose significantly improved the signs and symptoms of active SLE, with a high-resolution rate of 67% in SLEDAI-2K arthritis or rash, and showed a safety profile consistent with previous studies into baricitinib to treat RA. The study focused on specific organ manifestations, which benefited patients treated with baricitinib with rash and arthritis. So far, only one study has focused on the potential efficacy of baricitinib in SS. In that study, Aota et al. demonstrated baricitinib suppressed IFN-γ-induced CXCL10 expression in human salivary gland ductal cells and suggested its potential for the treatment of SS. Based on these, we thought that baricitinib might have therapeutic benefit in patients with pSS.

We plan to explore the efficacy and safety of baricitinib in patients with pSS in this single-center, prospective, open label, 24-weeks pilot study. We plan to enroll 11 patients diagnosed as active pSS in Peking Union Medical College Hospital, Beijing, China. They will be treated with baricitinib 2mg once a day for 24 weeks. We'll evaluate the disease activity mainly by ESSDAI and ESSPRI score. And we'll also record the adverse reactions. The primary endpoint of the study is the change of ESSDAI score at 12 weeks. The secondary endpoints include: the minimal clinically important improvement (MCII) of ESSDAI, which was defined as an improvement of ESSDAI of at least three points; the change of ESSDAI score at 24 weeks; the change of ESSPRI and PGA score at 12 and 24 weeks; and remissions of organ involvement at 12 and 24 weeks. The main inclusion criteria include: (1) ≥18 years old, (2) fulfill the criteria of the 2016 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification for primary SS, (3) with moderate or high activity of SS, which was defined as EULAR primary SS disease activity index (ESSDAI) ≥5, and (4) with serological activity defined as elevated C-reactive protein, erythrocyte sedimentation rate (ESR), and/or immunoglobulin G (IgG) level (excluding acute and chronic infection and other factors). The main exclusion criteria include: (1) patients diagnosed with an active central nervous system disease or dysfunction of a major organ (heart, liver, kidney); (2) pregnant or lactating women; (3) current severe infections; and (5) undergoing glucocorticoids or immunosuppressants treatment with stable dosage for less than 12 weeks.

DETAILED DESCRIPTION:
Baseline information included demographics, SS duration, clinical manifestations, laboratory parameters, current medications, and disease activity. Laboratory tests, including complete blood counts, urinalysis, liver and renal function tests, ESR, and IgG test were performed at each visit. Disease activity was assessed using the ESSDAI, EULAR primary SS patient reported index (ESSPRI), and physician global assessment (PGA) scores. Patients were followed up at 3 and 6 months after the initiation of baricitinib treatment. The concomitant medications including steroids and immunosuppressants were not changed during the study.

Response to treatment, or minimal clinically important improvement (MCII), was defined as an improvement of ESSDAI of at least three points23. Remissions of arthritis, cutaneous involvement, and hematological involvement were defined as no points earned in the corresponding items of the ESSDAI scoring system. The improvement of interstitial lung disease (ILD) was determined by evaluating the patient symptoms and radiographic changes in the pulmonary high-resolution computed tomography (HRCT) scan.

ELIGIBILITY:
Inclusion Criteria:

1. fulfill the criteria of the 2016 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification for primary SS
2. with moderate or high activity of SS, which was defined as EULAR primary SS disease activity index (ESSDAI) ≥5
3. with serological activity defined as elevated C-reactive protein, erythrocyte sedimentation rate (ESR), and/or immunoglobulin G (IgG) level (excluding acute and chronic infection and other factors)

Exclusion Criteria:

1. patients diagnosed with an active central nervous system disease or dysfunction of a major organ (heart, liver, kidney)
2. pregnant or lactating women
3. current severe infections
4. undergoing glucocorticoids or immunosuppressants treatment with stable dosage for less than 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
ESSDAI | 12 weeks
  the change of ESSDAI score at 12 weeks

SECONDARY OUTCOMES:
MCII of ESSDAI | 12 and 24 weeks
  Minimal clinically important improvement (MCII), defined as an improvement of ESSDAI of at least three points.
ESSDAI | 24 weeks
  the change of ESSDAI score at 24 weeks
ESSPRI | 12 and 24 weeks
  the change of ESSPRI score at 12 and 24 weeks
PGA | 12 and 24 weeks
  the change of PGA score at 12 and 24 weeks
remissions of organ involvement | 12 and 24 weeks
  Remissions of arthritis, cutaneous involvement, and hematological involvement were defined as no points earned in the corresponding items of the ESSDAI scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Leng, Dr., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years after article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to lengxm@gmail.com. To gain access, data requestors will need to sign a data access agreement.